CLINICAL TRIAL: NCT07301996
Title: Randomized Phase II Study to Evaluate Efficacy of Web-based Patient-reported Outcome (PRO) Application in Solid Cancer Patients
Acronym: Mobile PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sook Ryun Park, Associated Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0716; CB-2017-B-2 (Other Grant/Funding Number: 2017 Cancer Research Support Project of the Korea Foundation for Cancer Research)
Record Dates: First submitted 2025-11-30; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Solid Cancer
Keywords: Patient reported outcome

STUDY DESIGN:
Intervention Model Description: The intervention lasted 12 weeks. Patients in the Mobile PRO group received instruction on symptom reporting and were asked to submit reports at baseline and at least once before each outpatient visit. Treating oncologist reviewed Mobile PRO entries during clinic visits and used the information in clinical decision-making; no automated alerts or additional staff-based interventions were implemented.
  Usual-care patients did not use Mobile PRO; symptoms were assessed verbally during routine outpatient visits. AEs in both groups were graded using NCI-CTCAE version 5.0. All patients received chemotherapy according to institutional practice, including guideline-based antiemetic prophylaxis. Survival follow-up was conducted every 3 months after the 12-week intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile PRO (Experimental): Mobile PRO group. Patients in the Mobile PRO group received instruction on symptom reporting and were asked to submit reports at baseline and at least once before each outpatient visit. Treating oncologist reviewed Mobile PRO entries during clinic visits and used the information in clinical decision-making; no automated alerts or additional staff-based interventions were implemented.
  Interventions: Device: Mobile PRO
- Control (Sham Comparator): Usual group Usual-care patients did not use Mobile PRO; symptoms were assessed verbally during routine outpatient visits. AEs in both groups were graded using NCI-CTCAE version 5.0. All patients received chemotherapy according to institutional practice, including guideline-based antiemetic prophylaxis.
  Interventions: Other: usual care

INTERVENTIONS:
Device: Mobile PRO — Patients in the Mobile PRO group received instruction on symptom reporting and were asked to submit reports at baseline and at least once before each outpatient visit. Treating oncologist reviewed Mobile PRO entries during clinic visits and used the information in clinical decision-making; no automated alerts or additional staff-based interventions were implemented.
  Arms: Mobile PRO
Other: usual care — Usual-care patients did not use Mobile PRO; symptoms were assessed verbally during routine outpatient visits. AEs in both groups were graded using NCI-CTCAE version 5.0. All patients received chemotherapy according to institutional practice, including guideline-based antiemetic prophylaxis.
  Arms: Control

SUMMARY:
This is a single-center, open-label, Phase 2 study to evaluate the feasibility of a mobile PRO and its efficacy in reducing unplanned healthcare utilization (unplanned outpatient visits, emergency department visits, and hospitalizations).

DETAILED DESCRIPTION:
The intervention lasted 12 weeks. Patients in the Mobile PRO group received instruction on symptom reporting and were asked to submit reports at baseline and at least once before each outpatient visit. Treating oncologist reviewed Mobile PRO entries during clinic visits and used the information in clinical decision-making; no automated alerts or additional staff-based interventions were implemented.

Usual-care patients did not use Mobile PRO; symptoms were assessed verbally during routine outpatient visits. AEs in both groups were graded using NCI-CTCAE version 5.0. All patients received chemotherapy according to institutional practice, including guideline-based antiemetic prophylaxis. Survival follow-up was conducted every 3 months after the 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 years old
* Histologically or cytologically confirmed solid cancer (clinical diagnosis accepted for hepatocellular carcinoma per the American Association for the Study of Liver Disease guidelines)
* Receiving systemic therapy (cytotoxic, immunotherapy, targeted therapy, or combinations) as monotherapy or concurrent chemoradiotherapy
* Able to use a smartphone or tablet independently or with caregiver assistance.

Exclusion Criteria:

* Receiving third-line or later palliative systemic therapy
* Inability to understand PROM content.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Rate of unplanned healthcare utilization per patient | 12-week intervention period
  the composite of unplanned outpatient visits, emergency departments, visits, or hospitalizations.

SECONDARY OUTCOMES:
Impact on health-related QoL (HRQoL) | 12-week intervention period
  HRQoL was measured using the Korean version of EQ-5D-5L at baseline and 12 weeks, with index values derived from the Korean valuation set. For secondary analyses, EQ-5D-5L dimensions were dichotomized as "no problems" (Level 1) versus "any problems" (Levels 2-5).
Progression-free survival | From the date of starting chemotherapy to the date of first documentation of progression or death (up to approximately 1 years)
  The time from the date of starting chemotherapy to the date of disease progression as per RECIST version 1.1 or death from any cause, whichever occurs first.
Overall survival | From the date of starting chemotherapy to the date of death (up to approximately 1 years)
  The time from the date of starting chemotherapy to the date of death from any cause, whichever occurs first.
The proportions of individual components of unplanned healthcare use | 12-week intervention period
  Unplanned healthcare use was defined by its components: outpatient visits, emergency department visits, and hospital admissions. This outcome specifically measured the proportions of these three components.

OTHER OUTCOMES:
The rate of supportive medication prescriptions | 12-week intervention period
  The rate of supportive medication prescriptions, including anti-emetics, anti-diarrheal agents, digestives, analgesics, pegylated G-CSF, anti-histamine, corticosteroids, constipation medications, and other medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No